CLINICAL TRIAL: NCT05744219
Title: Improved Recovery by Iron Following Surgery With Blood Loss, a Double-blind Multi-centre Randomized Controlled Phase III Drug Trial (the IRIS-trial)
Brief Title: Improved Recovery by Iron Following Surgery With Blood Loss, the IRIS-trial
Acronym: IRIS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jon Unosson (Other)
Responsible Party: Sponsor-Investigator, Jon Unosson, Principal Investigator, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRIS
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Surgery; Liver Metastases; Liver Cancer; Pancreas Cancer; Aortic Aneurysm
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms; Aortic Aneurysm | interventions — ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: At end of surgery, peri-operative blood loss is determined and if 400-4000 ml, the patient is randomised to iv Ferric Carboxymaltose 1000 mg or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The attending nurse at the postoperative ward will do the final preparation of study drug and thus be aware of which patient receives placebo or iv iron. As the Ferric Carboxymaltose solution is opaque, the study drug is kept concealed behind the patient. Most patients have amnesia of the first hours after general anaesthesia. This effect is more pronounced after long and complex surgery which is the case for all patients included in this trial. Blinding from the patent's perspective is therefore not expected to be a major concern. The personnel preparing the study drug and nurse at the postoperative ward does not participate in care beyond this point, ensuring blinding is maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Iv Iron (Experimental): Ferric Carboxymaltose, single dose, Intra venous 1000 mg in 100 ml 0.9% NaCl
  Interventions: Drug: Ferric carboxymaltose
- Placebo (Placebo Comparator): Placebo, single dose, Intra venous 0.9% NaCl 100 ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — Active drug
  Arms: Iv Iron
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate if iv iron formulation improve recovery after surgery with blood loss.

Post-operative anaemia is a common debilitating condition after major surgery due to a combination of preoperative iron deficiency anaemia (IDA) and per-operative blood loss. Median blood loss following hepatopancreatobiliary (HPB) and complex aortic surgery typically range between 500-1000 ml. Bioavailability of iron may be a rate limiting factor in erythropoiesis in anaemia secondary to blood loss. For the IRIS trial, it is hypothesized that intravenously (iv) administered Ferric Carboxymaltose after a per-operative blood loss of 400-4000 ml, improves post-operative recovery and reduces the RBC transfusion.

Patients scheduled for elective HPB surgery or complex aortic surgery will be screened for eligibility and recruited into the study.

By the end of the surgical procedure, if blood loss is estimated to 400-4000 ml, the patient is randomized 1:1 to iv 1000 mg Ferric Carboxymaltose or placebo.

The primary endpoint is a composite of death, number of RBC transfusions, post-operative severe anemia (Hb <80 g/L) and FACT-An Quality of life (QoL) five weeks after surgery, assessed by win ratio.

The trial will also examine effects on; a) levels of Hb; b) markers of erythropoiesis and iron bioavailability; c) post-operative complications; d) post-operative recovery; e) performance status; f) subgroups based on type of surgery and degree of anemia and iron deficiency; g) re-admissions; h) long term outcome based on patient medical records and i) how post-operative recovery differs between those with low (<400 ml), high (400-4000 ml) and very high (>4000 ml) per-operative blood loss.

Recruitment will continue until 338 patients are randomized or 304 have completed the five week follow up

The coordinating center of the trial is the Department of Surgery at Uppsala University Hospital. Participating sites are also Linköping University Hospital and Lund University Hospital, all in Sweden. Other sites may be added.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent
2. Male and female patients
3. Weight > 50 kg
4. > 18 years of age
5. Scheduled for complex aortic surgery, liver resection or pancreatic resection

Exclusion Criteria:

1. Short expected survival (less than six months)
2. Intra-venous iron therapy within one month prior to surgery
3. Severe anaemia (B-Hb <80 mg/L) prior to surgery
4. Contraindication to Ferric Carboxymaltose according to SmPC
5. Iron overloading disorder, i.e. hemochromatosis
6. Risk of small for size future liver remnant
7. Pre-operative renal replacement therapy
8. Enrolled in another drug or medical device study within 30 days prior to enrolment of the current study
9. Another planned major surgical procedure before the five week follow up
10. Unsuitable for inclusion according to the investigator
11. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Recovery after iv Iron | Five weeks
  To examine if 1000 mg iv Ferric Carboxymaltose administered immediately following hepatic or pancreatic resection or complex aortic surgery with 400 - 4000 ml perioperative blood loss affect a composite of death, number of RBC transfusions, prevalence of post-operative severe anaemia (Hb < 80 g/L) and change in FACT-An QoL questionnaire score at five weeks after surgery compared to pre-operative baseline score. The composite endpoint is assessed by win ratio in the following order: Alive at five weeks (yes/no); number of RBC transfusions from surgery until five weeks; severe anaemia with Hb <80 g/L any time after surgery until five weeks (yes/no); FACT-An score (score at five weeks minus score at baseline)

SECONDARY OUTCOMES:
Hb | One to five weeks
  Assess if effects of the intervention are linked to increased post operative Hb (g/L)
Complications | One to five weeks
  To assess if the intervention reduce post operative complications measured by the comprehensive complication index
Recovery | One to five weeks
  To assess if the intervention affect recovery measured by the post operative morbidity survey
Performance status | Five weeks
  To assess if the intervention affect performance assessed by Karnofsky performance status

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala University Hospital, Uppsala, Sverige, Sweden

IPD SHARING:
Plan to Share IPD: No
May be available on request